CLINICAL TRIAL: NCT01990430
Title: Integrative Exercise and Life Style Intervention Increase Leisure Time Activity in Breast Cancer Patients.
Brief Title: Behavioural Changes in Breast Cancer Patients
Acronym: BHVBC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Politecnica de Madrid (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Puerta de Hierro University Hospital (Other); Hospital Universitario Madrid Sanchinarro (Other)
Responsible Party: Principal Investigator, Soraya Casla Barrio, Master, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: behaviourchanges
Record Dates: First submitted 2013-10-25; First posted 2013-11-21 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise Intervention (Experimental): The exercise program was designed and conducted by a qualified exercise physiologist with oncologic training. The exercise program consisted in a twice weekly supervised training program developed in a social framework. The sessions included instructions in training exercises, as well as included time to speak about their fears and doubts with other patients, who were in the same situation.
  The nutrition program consisted of three theoretical and practice classes, where specific terms of nutrition and diet were explained. Teachers did not promote avoiding any group of aliments and a Mediterranean diet was encouraged to be followed.
  Interventions: Behavioral: Exercise Intervention
- Control (No Intervention): Patients will be asked to maintain their usual life style, without special changes

INTERVENTIONS:
Behavioral: Exercise Intervention — Intervention: The sessions included instructions in training exercises, as well as included time to speak about their fears and doubts with other patients, who were in the same situation. The intervention lasted 12 weeks (24 sessions). The training intensity was progressively increased from 65% to 85% of heart rate with control by a POLAR FT7 heart rate monitor for aerobic activities, and by 8-15 repetitions in 2-3 sets for the strength activities. Exercise intensity was prescribed using Karvonen equation.
  The nutrition program consisted of three theoretical and practice classes. The first class explained the different groups of nutrients, their functions in the organism and for which group of aliments these can be obtained. The second class was a practical class about how to interpret food labels and relating measurements of food portions with recommendations for a healthy diet. Final session spoke about the ten best and the ten worst aliments, which prevent and promote cancer.
  Other Names: Active Life Style
  Arms: Exercise Intervention

SUMMARY:
Exercise training has been established as a feasible and safe intervention during or after neoplastic treatment in breast cancer patients. Numerous studies have shown that exercise can prevent and control various treatment-related side effects including functional limitation, physical capacity, anxiety and sleep disturbance. In the long-term, an active life style has been demonstrated to increase survival in women, who maintain a moderate level of exercise per week (30 or 75 minutes of brisk walking 5 days per week).

Specifically, active breast cancer survivors have a 51-85% lower cancer specific mortality and 33-82% lower all cause of mortality. But despite this, most breast cancer patients reduce their physical activity levels during and after cancer treatment. In 2010, a roundtable meeting of American College of Sport Medicine published guidelines for cancer survivors, defining that the recommended amount of exercise was 150 minutes per week of aerobic exercise of moderate-intensity and 2 or 3 days per week of strength training that included exercise for major muscle groups. But only 30-47% of breast cancer survivors follow these exercise recommendations.

In most clinical settings, information by the oncologist to keep physical active is part of the recommendation. Yet some breast cancer patients find it difficult to begin or maintain the minimal activity levels recommended by the experts. A typical obstacle includes lack of directions from experts, which can assure the safety and feasibility of the exercise that they perform. Moreover, important personal aspects can have major influence on the exercise preference, including certain food choice and dietary intakes, education level or the preference of a face-to-face exercise counseling by a professional.

A cancer diagnosis is recognized as "teachable moment", where patients are particularly motivated for lifestyle changes. So it is important to approach the patients with adequate interventions that consider the different needs in order to get a healthier behavior among the breast cancer patients.

Taking this into account, the hypothesis of this pilot project is that a guided integrated group exercise program, which includes an educational program on healthy life style, will increase the adherence of breast cancer survivors to exercise and a healthy diet. Therefore the aim of this pilot study was to investigate if a comprehensive and specific group exercise program, which includes dietary and exercise information, could increase leisure-time exercise in women with breast cancer.

DETAILED DESCRIPTION:
This study will be performed as a collaboration between Technical University of Madrid (UPM), Spanish Group of Cancer Patients (GEPAC), Hospital General Universitario Gregorio Marañón, Hospital Universitario Puerta de Hierr y Hospital de Sanchinarro-Madrid del Norte. The project will be carried out at the facilities of the Physical Activity and Sport Science Institute (INEF) and has been approved by the Ethical Committee of the UPM. A single arm pilot project with pre-post test has been designed.

Intervention The exercise program was designed and conducted by a qualified exercise physiologist with oncologic training. The exercise program consisted in a twice weekly supervised training program developed in a social framework. The sessions included instructions in training exercises, as well as included time to speak about their fears and doubts with other patients, who were in the same situation. The intervention lasted 12 weeks (24 sessions). The training intensity was progressively increased from 65% to 85% of heart rate with control by a POLAR FT7 heart rate monitor for aerobic activities, and by 8-15 repetitions in 2-3 sets for the strength activities. Exercise intensity was prescribed using Karvonen equation.

Every supervised session had the same structure and a duration of 60 minutes. American College Sport Medicine (ACSM) Guidelines for Cancer Patients were followed for the session design. The first 10 minutes was a dynamic warm up combining different ways of movement around the class and articular movements. Next part consisted in aerobic exercise, where the principal aim was to practice exercises that increased the participant's functional capacity with music-based activities such as aerobic, box-dance or global strength circuits without external resistance. Followed by upper-limbs strength exercises with elastic bands to improve strength and increase arm lean mass, focusing on chest and dorsal exercises. The last part was whole-body stretching exercises to improve joint mobility and muscle flexibility of upper body limbs, and general muscle relaxation after training.

The exercise program was complemented with theoretical classes about exercise and nutrition. One class of exercise prescription was held after two months of intervention. The patients were taught about the minimum of exercise recommended and about which activities they could do and how to adapt them depending on their own situations.

The nutrition program consisted of three theoretical and practice classes, where specific terms of nutrition and diet were explained. The first class explained the different groups of nutrients, their functions in the organism and for which group of aliments these can be obtained. The second class was a practical class about how to interpret food labels and relating measurements of food portions with recommendations for a healthy diet. Final session spoke about the ten best and the ten worst aliments, which prevent and promote cancer. Teachers did not promote avoiding any group of aliments and a Mediterranean diet was encouraged to be followed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Older than 18 years and younger than 75.
* Breast cancer diagnosed confirmed stage I-IIIA.
* Randomized disposition.
* Minimum of 45 days and maximum of 36 months after finishing treatments (chemotherapy and radiotherapy).
* 0-1 in Eastern Cooperative Oncology Group (ECOG) scale (present the ability to walk briskly)
* Oncologist approval.
* Informed Consent signed.
* Comunidad Autónoma de Madrid inhabitant.

Exclusion Criteria:

* Metastasis presence
* Serious medical risk such as unstable cardiac condition or severe pulmonary disease and anticoagulants treatments.
* Oncology or primary care approval who verified the medical risk exclusion criteria.
* ECOG > 1
* Pregnant

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Patients Quality of Life Questionnaire and Exercise Leisure-time Questionnaire | Changes from baseline at 12 weeks
  Combined primary objective has been elected. Both of them have to be positive. FACT-B and Godin Leisure-Time Exercise Questionnaire have been chosen as validated instruments to assess primary variables

SECONDARY OUTCOMES:
Fatigue Questionnaire | Changes from baseline at 12 weeks
  Fact-Fatigue (FACT-F) is the instrument chose to assess the variable
Depression Questionnaire | Change from baseline at 12 weeks
  Center of Epidemiologic Studies Depression Scale (CES-D scale) is the validated questioner chose to assess this variable

OTHER OUTCOMES:
Physical Capacity | Change from baseline at 12 weeks
  A maximal oxigen consumption (VO2) test will be used to assess this variable
Maximal Strength | Change from baseline at 12 weeks
  A 1 maximal repetition will be used to assess this variable

CONTACTS AND LOCATIONS:
Overall Officials: Javier Sampedro, Proffesor, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Faculty of Physical Activity and Sport Science, Madrid, Madrid, Spain

REFERENCES:
- [Background] Irwin ML, Crumley D, McTiernan A, Bernstein L, Baumgartner R, Gilliland FD, Kriska A, Ballard-Barbash R. Physical activity levels before and after a diagnosis of breast carcinoma: the Health, Eating, Activity, and Lifestyle (HEAL) study. Cancer. 2003 Apr 1;97(7):1746-57. doi: 10.1002/cncr.11227. PMID 12655532
- [Background] Mishra SI, Scherer RW, Geigle PM, Berlanstein DR, Topaloglu O, Gotay CC, Snyder C. Exercise interventions on health-related quality of life for cancer survivors. Cochrane Database Syst Rev. 2012 Aug 15;2012(8):CD007566. doi: 10.1002/14651858.CD007566.pub2. PMID 22895961
- [Background] Jones LW, Alfano CM. Exercise-oncology research: past, present, and future. Acta Oncol. 2013 Feb;52(2):195-215. doi: 10.3109/0284186X.2012.742564. Epub 2012 Dec 17. PMID 23244677
- [Background] Holmes MD, Chen WY, Feskanich D, Kroenke CH, Colditz GA. Physical activity and survival after breast cancer diagnosis. JAMA. 2005 May 25;293(20):2479-86. doi: 10.1001/jama.293.20.2479. PMID 15914748
- [Background] Betof AS, Dewhirst MW, Jones LW. Effects and potential mechanisms of exercise training on cancer progression: a translational perspective. Brain Behav Immun. 2013 Mar;30 Suppl(0):S75-87. doi: 10.1016/j.bbi.2012.05.001. Epub 2012 May 17. PMID 22610066
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Irwin ML. Physical activity interventions for cancer survivors. Br J Sports Med. 2009 Jan;43(1):32-8. doi: 10.1136/bjsm.2008.053843. Epub 2008 Oct 23. PMID 18948351
- [Background] Demark-Wahnefried W, Hars V, Conaway MR, Havlin K, Rimer BK, McElveen G, Winer EP. Reduced rates of metabolism and decreased physical activity in breast cancer patients receiving adjuvant chemotherapy. Am J Clin Nutr. 1997 May;65(5):1495-501. doi: 10.1093/ajcn/65.5.1495. PMID 9129482
- [Background] Hong S, Bardwell WA, Natarajan L, Flatt SW, Rock CL, Newman VA, Madlensky L, Mills PJ, Dimsdale JE, Thomson CA, Hajek RA, Chilton JA, Pierce JP. Correlates of physical activity level in breast cancer survivors participating in the Women's Healthy Eating and Living (WHEL) Study. Breast Cancer Res Treat. 2007 Jan;101(2):225-32. doi: 10.1007/s10549-006-9284-y. Epub 2006 Sep 21. PMID 17028988
- [Background] Jones LW, Courneya KS. Exercise counseling and programming preferences of cancer survivors. Cancer Pract. 2002 Jul-Aug;10(4):208-15. doi: 10.1046/j.1523-5394.2002.104003.x. PMID 12100105
- [Background] Blanchard CM, Courneya KS, Stein K; American Cancer Society's SCS-II. Cancer survivors' adherence to lifestyle behavior recommendations and associations with health-related quality of life: results from the American Cancer Society's SCS-II. J Clin Oncol. 2008 May 1;26(13):2198-204. doi: 10.1200/JCO.2007.14.6217. PMID 18445845
- [Background] Befort CA, Klemp JR, Austin HL, Perri MG, Schmitz KH, Sullivan DK, Fabian CJ. Outcomes of a weight loss intervention among rural breast cancer survivors. Breast Cancer Res Treat. 2012 Apr;132(2):631-9. doi: 10.1007/s10549-011-1922-3. Epub 2011 Dec 25. PMID 22198470
- [Background] Hayes SC, Johansson K, Stout NL, Prosnitz R, Armer JM, Gabram S, Schmitz KH. Upper-body morbidity after breast cancer: incidence and evidence for evaluation, prevention, and management within a prospective surveillance model of care. Cancer. 2012 Apr 15;118(8 Suppl):2237-49. doi: 10.1002/cncr.27467. PMID 22488698
- [Background] Giacosa A, Barale R, Bavaresco L, Gatenby P, Gerbi V, Janssens J, Johnston B, Kas K, La Vecchia C, Mainguet P, Morazzoni P, Negri E, Pelucchi C, Pezzotti M, Rondanelli M. Cancer prevention in Europe: the Mediterranean diet as a protective choice. Eur J Cancer Prev. 2013 Jan;22(1):90-5. doi: 10.1097/CEJ.0b013e328354d2d7. PMID 22644232
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Valenti M, Porzio G, Aielli F, Verna L, Cannita K, Manno R, Masedu F, Marchetti P, Ficorella C. Physical exercise and quality of life in breast cancer survivors. Int J Med Sci. 2008 Jan 15;5(1):24-8. doi: 10.7150/ijms.5.24. PMID 18219372
- [Background] Eyigor S, Karapolat H, Yesil H, Uslu R, Durmaz B. Effects of pilates exercises on functional capacity, flexibility, fatigue, depression and quality of life in female breast cancer patients: a randomized controlled study. Eur J Phys Rehabil Med. 2010 Dec;46(4):481-7. PMID 21224783
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] van Waart H, Stuiver MM, van Harten WH, Sonke GS, Aaronson NK. Design of the Physical exercise during Adjuvant Chemotherapy Effectiveness Study (PACES): a randomized controlled trial to evaluate effectiveness and cost-effectiveness of physical exercise in improving physical fitness and reducing fatigue. BMC Cancer. 2010 Dec 7;10:673. doi: 10.1186/1471-2407-10-673. PMID 21138561
- [Background] Delgado-Sanz MC, Garcia-Mendizabal MJ, Pollan M, Forjaz MJ, Lopez-Abente G, Aragones N, Perez-Gomez B. Heath-related quality of life in Spanish breast cancer patients: a systematic review. Health Qual Life Outcomes. 2011 Jan 14;9:3. doi: 10.1186/1477-7525-9-3. PMID 21235770
- [Background] Brown JC, Huedo-Medina TB, Pescatello LS, Ryan SM, Pescatello SM, Moker E, LaCroix JM, Ferrer RA, Johnson BT. The efficacy of exercise in reducing depressive symptoms among cancer survivors: a meta-analysis. PLoS One. 2012;7(1):e30955. doi: 10.1371/journal.pone.0030955. Epub 2012 Jan 27. PMID 22303474